CLINICAL TRIAL: NCT00261950
Title: Bone Histomorphometry Assessment For Dialysis Patients With Secondary Hyperparathyroidism of End Stage Renal Disease
Brief Title: Bone Biopsy Study For Dialysis Patients With Secondary Hyperparathyroidism of End Stage Renal Disease
Acronym: BONAFIDE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050104; BONAFIDE Study (Other: Amgen); IND #56,010 (Other: Food and Drug Administration)
Record Dates: First submitted 2005-12-02; First posted 2005-12-06 (Estimated); Results first posted 2013-12-04 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-06

CONDITIONS: Secondary Hyperparathyroidism
Keywords: Cinacalcet HCl, Cinacalcet, Amgen (AMG) 073, Sensipar, Mimpara, Calcimimetic
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — Cinacalcet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cinacalcet (Experimental): All subjects were enrolled into the single arm to receive Cinacalcet. There was no comparator arm.
  Interventions: Drug: Sensipar (Cinacalcet HCl)

INTERVENTIONS:
Drug: Sensipar (Cinacalcet HCl) — All enrolled subjects receive study medication at a starting dose of 30 mg cinacalcet once daily beginning on day 1. Possible sequential doses are 30 mg, 60mg, 90mg, 120mg, 180 mg taken once daily. During the study, dose adjustment (dose increase/decrease/withholding) is based upon iPTH, serum calcium, and subject safety information. Subjects swallowed tablets whole without biting or chewing. Subjects were dispensed investigational product every 4 weeks starting from Day 1 through to Week 48.

SUMMARY:
The purpose of this study is to evaluate the effects of cinacalcet on markers of bone turnover in patients with kidney disease who are receiving dialysis.

DETAILED DESCRIPTION:
Secondary hyperparathyroidism (HPT) is common in people with end stage renal disease (kidney disease). Patients with secondary HPT often have enlarged parathyroid glands in the neck and as a result often have elevated parathyroid hormone (PTH) levels . Patients with secondary HPT may have bone disease (osteodystrophy). Cinacalcet has been used to decrease PTH levels in patients with secondary HPT. Patients with secondary HPT may have bone disease (osteodystrophy). This bone disease may cause bone pain, fractures, and poor formation of red blood cells. The purpose of this study is to evaluate effects of cinacalcet on markers of bone turnover in patients with kidney disease who are receiving dialysis.

ELIGIBILITY:
Inclusion Criteria: Subjects will be eligible for the study if they meet all of the following criteria:

* One Intact Parathyroid Hormone (iPTH) determination obtained from the central laboratory must be >/= 300 pg/mL.
* One serum calcium determination obtained from the central laboratory must be >/= 8.4 mg/dL (2.1 mmol/L).
* One Bone Alkaline Phosphatase (BALP) determination obtained from the central laboratory must be >/= 20.9 ng/mL.
* Positive histologic confirmation of high bone turnover disease as assessed by the central bone histology center.
* Treated with dialysis >/= 1 month before the date of informed consent.

Exclusion Criteria: Subjects will be ineligible for the study if they:

* Have an unstable medical condition in the judgment of the investigator.
* Are pregnant or nursing women.
* Had a parathyroidectomy in the 3 months before the date of informed consent.
* For subjects prescribed vitamin D, have received vitamin D therapy for less than 30 days before day 1 or required a change in vitamin D brand or dose level within 30 days before day 1.
* Ever received therapy with Sensipar®/Mimpara®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2006-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (52):
- United States (16):
  - Research Site, Phoenix, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Denver, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Evanston, Illinois
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, Teaneck, New Jersey
  - Research Site, Flushing, New York
  - Research Site, Great Neck, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Allentown, Pennsylvania
  - Research Site, Houston, Texas
- Belgium (4):
  - Research Site, Antwerp
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Liège
- Czechia (2):
  - Research Site, Hradec Králové
  - Research Site, Prague
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
- Italy (8):
  - Research Site, Avellino
  - Research Site, Cremona
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Ortona CH
  - Research Site, Ostia RM
  - Research Site, Roma
  - Research Site, Roma (RM)
- Research Site, Skopje, North Macedonia
- Poland (3):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Wroclaw
- Portugal (6):
  - Research Site, Porto, PR
  - Research Site, Almada
  - Research Site, Estoril
  - Research Site, Guimarães
  - Research Site, Porto
  - Research Site, Vila Franca de Xira
- Spain (4):
  - Research Site, Santander, Cantabria
  - Research Site, Barcelona, CataluÃ±a
  - Research Site, AlcorcÃ³n, Madrid
  - Research Site, Madrid, Madrid
- Research Site, Zurich, Switzerland
- Research Site, Izmir, Turkey (Türkiye)
- Research Site, Manchester, United Kingdom

REFERENCES:
- [Background] TBD.BONAFIDE Baseline/Primary Results.Journal-004521;
- [Background] Behets GJ, Spasovski G, Sterling LR, Goodman WG, Spiegel DM, De Broe ME, D'Haese PC. Bone histomorphometry before and after long-term treatment with cinacalcet in dialysis patients with secondary hyperparathyroidism. Kidney Int. 2015 Apr;87(4):846-56. doi: 10.1038/ki.2014.349. Epub 2014 Oct 22. PMID 25337774
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: May 22 2006 is study initiation date and 13 May 2011 is study completion date.
Groups:
- Cinacalcet: cinacalcet hydrochloride. Participants received a starting dose of 30 mg cinacalcet daily (QD). Dose adjustments were based upon repeated measurements of intact parathyroid hormone, calcium serum concentrations, and participant safety information.
Period: Overall Study
Arm/Group | Cinacalcet
Started | 110
Completed | 84
Not Completed | 26
Not completed — Lost to Follow-up | 2
Not completed — Death | 6
Not completed — Withdrawal by Subject | 5
Not completed — Other | 1
Not completed — Physician Decision | 1
Not completed — Protocol specified Criteria | 11

BASELINE CHARACTERISTICS:
Arm/Group | Cinacalcet
Number analyzed (Participants) | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 70
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 91
  Black | 10
  Other | 9

OUTCOME MEASURES:

1. Secondary Outcome: Percent Change From Baseline in Serum Calcium During the Efficacy Assessment Phase (EAP)
Time Frame: Baseline to weeks 40-52
Population: Enrolled subjects with serum calcium during the Efficacy Assessment Phase (EAP)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Cinacalcet
Number analyzed (Participants) | 74
percent change | -6.5 (1.1)

2. Secondary Outcome: Percent Change From Baseline in Serum Phosphorus During the Efficacy Assessment Phase (EAP)
Time Frame: Baseline to weeks 40-52
Population: Enrolled subjects with serum phosphorus during the Efficacy Assessment Phase (EAP)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Cinacalcet
Number analyzed (Participants) | 74
percent change | -1.1 (2.9)

3. Secondary Outcome: Percent Change From Baseline in Ca x P During the Efficacy Assessment Phase (EAP)
Time Frame: Baseline to weeks 40-52
Population: Enrolled subjects with Ca x P during the Efficacy Assessment Phase (EAP)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Cinacalcet
Number analyzed (Participants) | 74
percent change | -6.9 (3.1)

4. Secondary Outcome: Percent Change From Baseline in Bone Specific Alkaline Phosphatase (BALP) at Week 52
Time Frame: Baseline to week 52
Population: Enrolled subjects with BALP at week 52
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Cinacalcet
Number analyzed (Participants) | 73
percent change | 6.6 (12.7)

5. Secondary Outcome: Percent Change From Baseline in N - Telopeptide (NTx) at Week 52
Time Frame: Baseline to week 52
Population: Enrolled subjects with NTx at week 52
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Cinacalcet
Number analyzed (Participants) | 72
percent change | -14.0 (14.7)

6. Secondary Outcome: Percent Change From Baseline in Parathyroid Hormone (PTH) During the Efficacy Assessment Phase (EAP)
Time Frame: Baseline to weeks 40-52
Population: Enrolled subjects with PTH during the Efficacy Assessment Phase (EAP)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Cinacalcet
Number analyzed (Participants) | 74
percent change | -41.6 (4.4)

7. Primary Outcome: Change From Baseline to End of Study in Bone Formation Rate (BFR)
Time Frame: Baseline to week 52
Population: Enrolled subjects with bone biopsy at week 52
Measure: Mean (Standard Error); unit: μm^2/mm^2/day
Arm/Group | Cinacalcet
Number analyzed (Participants) | 77
μm^2/mm^2/day | -488 (73)

8. Secondary Outcome: Change From Baseline to End of Study in Osteoblast Perimeter (Osteoblast Perimeter/Osteoid Perimeter)
Description: Osteoblast Perimeter was calculated as "Osteoblast Perimeter/Osteoid Perimeter * 100"
Time Frame: Baseline to week 52
Population: Enrolled subjects with Osteoblast Perimeter at week 52
Measure: Mean (Standard Error); unit: percentage of osteoid perimeter
Arm/Group | Cinacalcet
Number analyzed (Participants) | 77
percentage of osteoid perimeter | -4.3 (1.4)

9. Secondary Outcome: Change From Baseline to End of Study in Osteoclast Perimeter (Osteoclast Perimeter/Eroded Perimeter)
Description: Osteoclast Perimeter was calculated as "Osteoclast Perimeter/Eroded Perimeter * 100"
Time Frame: Baseline to week 52
Population: Enrolled subjects with Osteoclast Perimeter at week 52
Measure: Mean (Standard Error); unit: percentage of eroded perimeter
Arm/Group | Cinacalcet
Number analyzed (Participants) | 77
percentage of eroded perimeter | -2.7 (1.5)

10. Secondary Outcome: Change in Categorization From Baseline to End of Study in Fibrosis Area/Tissue Area
Description: Categorisation at each timepoint was based on fibrosis area as a percentage of tissue area (Fibrosis Area/Tissue Area * 100)
Time Frame: Baseline to week 52
Population: Enrolled subjects with Fibrosis Area/Tissue Area at week 52
Measure: Number; unit: participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 77
participants
  Baseline 0% End of Study 0% | 3
  Baseline 0% End of Study 1-5% | 3
  Baseline 0% End of Study 6-10% | 0
  Baseline 0% End of Study 11-25% | 0
  Baseline 0% End of Study ≥ 26% | 0
  Baseline 1-5% End of Study 0% | 17
  Baseline 1-5% End of Study 1-5% | 31
  Baseline 1-5% End of Study 6-10% | 2
  Baseline 1-5% End of Study 11-25% | 0
  Baseline 1-5% End of Study ≥ 26% | 0
  Baseline 6-10% End of Study 0% | 4
  Baseline 6-10% End of Study 1-5% | 7
  Baseline 6-10%% End of Study 6-10% | 5
  Baseline 6-10% End of Study 11-25% | 2
  Baseline 6-10% End of Study ≥ 26% | 0
  Baseline 11-25% End of Study 0% | 0
  Baseline 11-25% End of Study 1-5% | 0
  Baseline 11-25% End of Study 6-10% | 1
  Baseline 11-25% End of Study 11-25% | 0
  Baseline 11-25% End of Study ≥ 26% | 0
  Baseline ≥ 26% End of Study 0% | 0
  Baseline ≥ 26% End of Study 1-5% | 1
  Baseline ≥ 26% End of Study 6-10% | 1
  Baseline ≥ 26% End of Study 11-25% | 0
  Baseline ≥ 26% End of Study ≥ 26% | 0

11. Secondary Outcome: Change From Baseline to End of Study in Eroded Perimeter/Bone Perimeter
Description: Eroded Perimeter/Bone Perimeter was calculated as "Eroded Perimeter/Bone Perimeter * 100"
Time Frame: Baseline to week 52
Population: Enrolled subjects with eroded perimeter/bone perimeter at week 52
Measure: Mean (Standard Error); unit: percentage of bone perimeter
Arm/Group | Cinacalcet
Number analyzed (Participants) | 77
percentage of bone perimeter | -3.4 (0.6)

12. Secondary Outcome: Percent Change From Baseline in Osteocalcin (OC) at Week 52
Time Frame: Baseline to week 52
Population: Enrolled subjects with osteocalcin (OC) at week 52
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Cinacalcet
Number analyzed (Participants) | 68
Percent change | -21.8 (6.2)

13. Secondary Outcome: Percent Change From Baseline in Tartrate Resistant Acid Phosphatase(TRAP) at Week 52
Time Frame: Baseline to week 52
Population: Enrolled subjects with TRAP at week 52
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Cinacalcet
Number analyzed (Participants) | 71
percent change | -3.8 (9.2)

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Cinacalcet
Serious Adverse Events (participants affected / at risk) | 45/110
Other Adverse Events (participants affected / at risk) | 84/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cinacalcet (N=110)
Anaemia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 2
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 3
Myocardial ischaemia (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Hyperparathyroidism secondary (Endocrine disorders) | 1
Diplopia (Eye disorders) | 1
Papilloedema (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 3
Death (General disorders) | 1
Facial pain (General disorders) | 1
Impaired healing (General disorders) | 1
Pyrexia (General disorders) | 2
Bile duct obstruction (Hepatobiliary disorders) | 1
Acinetobacter infection (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Breast abscess (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Escherichia bacteraemia (Infections and infestations) | 1
Escherichia infection (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Infected skin ulcer (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Sepsis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Blood pressure increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diabetic foot (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression suicidal (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Swelling face (Skin and subcutaneous tissue disorders) | 1
Arterial disorder (Vascular disorders) | 1
Arteriovenous fistula (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Intra-abdominal haemorrhage (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cinacalcet (N=110)
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 22
Dyspepsia (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 28
Vomiting (Gastrointestinal disorders) | 23
Oedema peripheral (General disorders) | 6
Pyrexia (General disorders) | 6
Bronchitis (Infections and infestations) | 8
Upper respiratory tract infection (Infections and infestations) | 6
Procedural pain (Injury, poisoning and procedural complications) | 8
Decreased appetite (Metabolism and nutrition disorders) | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Headache (Nervous system disorders) | 8
Insomnia (Psychiatric disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Hypertension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.